CLINICAL TRIAL: NCT05755724
Title: Remote Immersive Virtual Reality (RIVR) Teaching: Use in Ultrasound Guided Regional Anesthesia Procedural Skills Acquisition
Brief Title: Remote Immersive Virtual Reality Teaching:
Acronym: RIVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Ahtsham Niazi, Associate Professor, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 5424
Record Dates: First submitted 2023-02-11; First posted 2023-03-06 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Educational Problems; Acute Pain
Keywords: Regional Anesthesia; Education; Ultrasound
MeSH Terms: conditions — Acute Pain | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The study will be designed as a single-centre, prospective, double blinded, randomized (1:1) trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote immersive virtual reality group (3D) teaching (Experimental): Telesimulation using immersive VR technology. Briefly, students will have a 360° camera mounted to their head, which will broadcast their first-person perspective to their teachers. Teachers will be able to immerse themselves in the perspective of the trainee using a virtual reality HMD (Oculus Quest 2), which allows them to look around freely and view equipment, hand movements, etc. and offer instruction accordingly.
  Interventions: Other: 3-D Teaching
- Remote 2 D teaching (Placebo Comparator): Telesimulation using standard teleconferencing software and equipment including 2D computer monitors, webcams, and an ultrasound machine linked to a computer (enabling ultrasound images to be transmitted).
  Interventions: Other: 2-D Teaching

INTERVENTIONS:
Other: 3-D Teaching — Telesimulation using immersive VR technology. Briefly, students will have a 360° camera mounted to their head, which will broadcast their first-person perspective to their teachers. Teachers will be able to immerse themselves in the perspective of the trainee using a virtual reality HMD (Oculus Quest 2), which allows them to look around freely and view equipment, hand movements, etc. and offer instruction accordingly.
  Other Names: Remote immersive virtual reality group (3D) teaching
  Arms: Remote immersive virtual reality group (3D) teaching
Other: 2-D Teaching — Telesimulation using standard teleconferencing software and equipment including 2D computer monitors, webcams, and an ultrasound machine linked to a computer (enabling ultrasound images to be transmitted).
  Other Names: Remote 2 D Teaching
  Arms: Remote 2 D teaching

SUMMARY:
Patients in rural Canada face serious anesthesia care deficiencies relative to their counterparts in urban centers. Despite 18% of Canadians living in rural settings only 3.1% of medical specialists practice in rural areas. To provide equity in healthcare there is a need to develop a network where specialists in urban centers can provide training, coaching, and support to physicians in rural communities. Despite some work being done this is not possible for all specialists due to cost and travel. One potential solution to this problem is telesimulation, whereby telecommunication and simulation tools are used to provide training remotely. Simple, 2D telesimulation setups using webcams and computers have been used to teach remotely but problems with video displays and learner engagement have occurred leading to a need for more sophisticated telesimulation tools. Recently, virtual reality (VR) systems have been developed allowing the learner and teacher to immerse in a 3D computer-generated environment where they feel as if they are in the same room. We propose to see whether teaching ultrasound guided regional anesthesia (UGRA), a skill required by rural physicians, using 3D VR is better than teaching by 2D tele simulation.

DETAILED DESCRIPTION:
Introduction:

Ultrasound-guided regional anesthesia (UGRA) has many advantages over traditional regional anesthesia approaches; however, it requires the acquisition of several new technical and non-technical skills. Successful acquisition of these skills is relatively complex, and generally not achievable through didactic teaching alone, thus the majority of UGRA training takes place from expert-guided 'hands-on' teaching workshops. However, barriers such as travel time and associated costs limit attendance at these workshops, especially for physicians in remote and rural areas, increasing the inequality experienced by rural medicine patients and practitioners.

One potential solution to this problem is telesimulation, whereby telecommunication and simulation tools are used to provide training remotely. Indeed simple, 2D telesimulation setups using webcams and computers have been used to successfully teach UGRA in remote areas. More sophisticated telesimulation tools have recently been developed with elements of immersive virtual reality (VR), i.e., a 3D computer-generated world including sensory feedback that users can interact with. A simple and cost-effective immersive VR approach to telesimulation includes a 360° camera and a VR headset/head mounted display (HMD), which has the potential to immerse a teacher into the learner's environment, allowing the teacher to see the learner's movements and actions in the first person.

Recent advancements in VR technology have reduced costs and increased accessibility, and 360° VR video can benefit learning processes by boosting motivation and encouraging knowledge retention. Thus, the investigators propose to compare remote teaching of UGRA using Remote Immersive VR (RIVR) and 2D telesimulation teaching.

Purpose:

As highlighted in a recent report, patients, and healthcare practitioners in rural Canada face serious deficiencies relative to their counterparts in urban centres. Despite 18% of Canadians living in rural settings only 3.1% of medical specialists practice in rural areas. Thus, there is a strong need for teaching and mentorship among anesthetists in Canada's remote communities. This study will directly address two of the recommendations in this report by assessing coaching tools which can guide improvements in the clinical practice of rural physicians and by facilitating networks of care between urban specialists and rural centers.

By directly comparing two training methods, the investigators will also increase knowledge of telesimulation best practices and immersive VR as a training modality, potentially leading to better educational outcomes for students and ultimately to better clinical outcomes for patients. This is in alignment with the Sunnybrook Education Strategic Plan goal, to improve learner, teacher and patient experiences and outcomes through education research and scholarship.

Hypothesis:

The investigators hypothesize that telesimulation training through 3D RIVR will provide a more effective method of teaching UGRA than the use of 2D teleconferencing (i.e., using webcams and computer screens).

Study Objective:

To compare two telesimulation methods, 2D video and 3D RIVR, for remote teaching of UGRA.

Study Design:

The study will be designed as a single-centre, prospective, assessor blinded, randomized (1:1) trial.

Recruitment:

Advertisements for eligible participants will be sent via electronic and hard copy formats. These include emails via faculties/schools of medicine, hospital bulletin boards and student common rooms. In all approaches, advertisements will ask for volunteers for the study and will include details to contact a researcher via email or telephone.

Permission to access medical students will be sought via the faculties/schools of medicine, with the advertisement sent on researcher's behalf. Researchers will not be seeking access or retention of student email addresses.

A manual check of eligibility and exclusion criteria will be performed for all participants. An informed consent form (ICF) will be provided. After consenting to participate, all participants will be allocated a number and remain de-identified throughout the data collection process.

Intervention and Randomization:

Following ethics approval, 24 medical students from the University of Toronto, with no prior ultrasound experience, will be recruited to participate in this study. Students will be randomized (1:1) to receive remote UGRA instruction using either 2D telesimulation technology or 3D RIVR. Both groups will also use a simulation model on which needle insertion, needle alignment, target acquisition and injection of local anesthetic will be taught.

2D Group: Telesimulation using standard teleconferencing software and equipment including 2D computer monitors, webcams, and an ultrasound machine linked to a computer (enabling ultrasound images to be transmitted).

3D RIVR Group: Telesimulation using immersive VR technology. Briefly, students will have a 360° camera mounted to their head, which will broadcast their first-person perspective to their teachers. Teachers will be able to immerse themselves in the perspective of the trainee using a virtual reality HMD (Oculus Quest 2), which allows the teacher to look around freely and view equipment, hand movements, etc. and offer instruction accordingly.

Evaluation:

Prior to teaching, students in both groups will undergo a pretest using a validated, 22-item procedural checklist and a 9-item Global Rating Scale (GRS). After the pretest, the students will be provided with a PowerPoint presentation including basic knowledge of the ultrasound machine, the simulation model, and the UGRA procedure. Students will then be invited back after an hour and provided with a one-hour session of teaching on how to perform an ultrasound-guided nerve block by an instructor in another room via telesimulation (either 2D or 3D RIVR). After the session, students will be asked to undergo a posttest evaluation using the same GRS and checklist. The pretest and posttest will be recorded and assessed by two experts in UGRA who are blinded to the method of teaching. The two evaluators will score each participant independently and the scores will be averaged.

Study Outcomes:

Primary Outcome: Difference in scores from before (pretest) to after training (posttest) as assessed using a validated procedural checklist and Global Rating Scale (GRS) for assessment of UGRA.

Expected Outcome: The investigators expect to see greater improvements in pretest to posttest scores using 3D RIVR, relative to 2D telesimulation.

Secondary Outcomes: Time required to teach UGRA using each modality, qualitative assessment of teacher and student satisfaction for each modality, quality of teaching using each method (e.g., how well the teaching instructions were delivered and acted upon) as evaluated by two blinded assessors.

Expected Outcome: The investigators will identify additional advantages and potential barriers related to the use of 3D RIVR for remote telesimulation training of complex technical and non-technical skills, relative to 2D telesimulation.

Statistical Analysis:

Sample size calculation was performed based on the conservative assumption that participants will have an average percentage score of 60% (SD 20%) in the pretest, given their minimal training in ultrasound and lack of familiarity with UGRA. The analysis of the primary outcome (GRS and checklist) will be compared between groups using the paired sample t-test (two-sided, where P < 0.05 will be considered statistically significant). A score of 80% on the posttest will be chosen to represent a successful posttest score (i.e., significant improvement), as previously described. Based on Type I error of 0.05 and beta = 0.1, 11 participants per group (22 total) are required. The investigators aim to recruit 24 participants to compensate for any attrition during the study.

Impact:

The goal of this project is to identify the most effective way to remotely teach the complex skills required for UGRA procedures. This will allow specialist physicians working in large urban centres to share their knowledge more widely, and directly benefit physicians working in remote communities, by giving rural physicians access to expert teaching and mentorship. This, in turn, will increase access to specialist care for patients living in remote and rural communities, improving outcomes and allowing patients to access care where they live.

Furthermore, by providing evidence to support the use of 3D RIVR for teaching both technical and non-technical skills, the investigators will increase their knowledge related to the use of this novel technology and provide a proof-of-concept, which could be applied to other techniques and medical specialties.

ELIGIBILITY:
Inclusion Criteria:

* Participants are medical students from year 1 and 2

Exclusion Criteria:

* Participants with any prior exposure (workshop, lecture, tutorial, actual performance) of ultrasound guided procedures, including regional anesthesia.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Difference in scores from before (pretest) to after training (posttest) using an Assessment Checklist for Ultrasound-Guided Regional Anesthesia. | 15 minutes
  Difference in scores from before (pretest) to after training (posttest) will be assessed using a validated procedural checklist termed as the Assessment Checklist for Ultrasound-Guided Regional Anesthesia. The checklist has 22 items which will be graded as not performed (0 Marks), performed poorly (1 Mark), or performed well (2 Marks).
Difference in scores from before (pretest) to after training (posttest) using an Global Rating Scale (GRS) for assessment of Ultrasound Guided Regional Anesthesia. | 15 minutes
  Difference in scores from before (pretest) to after training (posttest) will be assessed using a validatedGlobal Rating Scale termed as the Global Rating Scale (GRS) for assessment of Ultrasound Guided Regional Anesthesia.The GRS has 9 items with a score of 1-5 for each item, with 1 correlating to a very poor performance and 5 correlating to a clearly superior performance.

SECONDARY OUTCOMES:
Qualitative assessment of teacher and student satisfaction for each modality | 10 minutes
  Satisfaction survey for both instructor and student consisting of seven questions with a five point scale looking at whether the teacher/participant Highly agrees, Somewhat agrees, is neutral, Somewhat disagrees and Highly disagrees.
Time required to teach UGRA using each modality | 10 minutes
  Time taken to teach

CONTACTS AND LOCATIONS:
Overall Officials: Ahtsham U Niazi, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada